CLINICAL TRIAL: NCT05319795
Title: Exploring the Efficacy of the Effortful Swallow Maneuver for Improving Swallowing in People With Parkinson Disease
Brief Title: Effortful Swallow Maneuver for Swallowing Impairment in People With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Catriona Steele, Scientist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPCR 21-5814
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Dysphagia
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: This is a prospective single arm case series treatment study involving a behavioral intervention (the Effortful Swallow Maneuver).
Masking Description: This is a single arm study. However, individuals responsible for rating the videofluoroscopy x-ray data to determine outcomes will be blinded to timepoint of evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effortful Swallow Maneuver (Experimental): Adults with a confirmed diagnosis of Parkinson Disease who have radiographically confirmed difficulties with timely airway protection and/or bolus clearance during swallowing. Individuals will complete a 4-week intervention program with two 30-minute sessions of Effortful Swallow (ES) practice daily, 5 days per week.
  Interventions: Behavioral: Effortful Swallow Maneuver

INTERVENTIONS:
Behavioral: Effortful Swallow Maneuver — Repeated practice of the Effortful Swallowing Maneuver generated by pushing the tongue with increased effort against the palate at the point of swallow initiation.

SUMMARY:
Context: Many people with Parkinson Disease (PwPD) experience swallowing difficulties, particularly with food/liquid going down the wrong way or remaining in the throat after swallowing. Prior studies suggest that exercise-based treatments targeting swallowing strength may be effective in reducing these difficulties.

Research question: Does an exercise-based treatment involving the effortful swallow maneuver improve swallowing function in PwPD?

Study plan: The investigators will study the effects of a four-week intensive swallowing rehabilitation program in PwPD, over a 2-year period.

DETAILED DESCRIPTION:
The investigators will study the effects of a four-week intensive swallowing rehabilitation program in PwPD, over a 2 year period. The program will involve daily practice of the effortful swallowing maneuver, with swallowing function assessed before and after the treatment program using videofluoroscopic x-rays.

Expected outcomes: In other populations, the effortful swallow has shown to address two mechanisms that are thought to underlie swallowing impairment in Parkinson Disease: slowness in achieving airway protection and weakness in muscles responsible for transporting food through the throat. The investigators expect that repeated practice of this maneuver by PwPD will lead to improved airway protection and improved clearance of residue from the throat.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* English-speaking
* Able to follow study instructions
* Neurologist confirmed diagnosis of PD
* Hoehn and Yahr scale score of 2 or 3
* Self-report of one or more swallowing or related symptoms:

  1. Difficulty with secretion management
  2. Coughing at the meal time
  3. Choking on food
  4. Respiratory infection in the past 6 months (other than COVID)

Exclusion Criteria:

* History of head and neck cancer
* Radical neck dissection (e.g. anterior cervical spine surgery) or neck/ oropharyngeal surgery (not excluded - tonsillectomy, adenoidectomy)
* Past medical history of any neurological disease other than PD (e.g. multiple sclerosis, amyotrophic lateral sclerosis, traumatic brain injury, stroke)
* Cognitive or receptive communication difficulties that preclude the participant's ability to follow study instructions provided in English. This will be determined by the participant's physician prior to referring them to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona M Steele, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Effortful Swallow Maneuver
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 70 [63 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Time-to-laryngeal-vestibule-closure Thin Liquids
Description: The time interval (in milliseconds) measured on a videofluoroscopic x-ray of swallowing between onset of the hyoid burst movement at the beginning of a swallow and achieving airway protection via closure of the laryngeal vestibule. The investigators will measure time-to-laryngeal-vestibule-closure across a series of 3 thin liquid swallows in videofluoroscopy. The participant's worst score (i.e. longest) across these 3 task repetitions will be recorded at each timepoint and the difference across timepoints will be calculated.
Time Frame: Post treatment (4 weeks) compared to pre-treatment baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
milliseconds | 0 (132)

2. Primary Outcome: Change in Penetration-Aspiration Scale Score Thin Liquids
Description: The Penetration-Aspiration Scale is an 8-point ordinal scale, measured on a videofluorosopic x-ray of swallowing, which documents the depth of any airway invasion events, and the subsequent response to airway invasion (Rosenbek et al., 1996). The scale ranges from a minimum score of 1 (no airway invasion) to a maximum score of 8 (entry of material below the true vocal folds with no response and no ejection). Higher scores are worse. The investigators will measure penetration-aspiration across a series of 3 thin liquid swallows in videofluoroscopy. The participant's worst score (i.e. highest) across these three task repetitions will be recorded at each timepoint and the difference across timepoints will be calculated.
Time Frame: Post treatment (4 weeks) compared to pre-treatment baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
score on a scale | 0 (1)

3. Primary Outcome: Change in Pharyngeal Area at Maximum Constriction Thin Liquids
Description: A videofluoroscopic measure of the degree of pharyngeal constriction during swallowing (i.e. maximum obliteration of the space in the pharynx). This measure is obtained from pixel-based measures of the unobliterated area of the pharynx on a lateral view x-ray image at the point of maximum constriction. The number of pixels is divided by an anatomical reference scalar defined by the squared length of the distance, in pixels, between the anterior inferior corners of the C2 and C4 cervical vertebrae on the same image. The investigators will measure pharyngeal area at maximum constriction across a series of 3 thin liquid swallows in videofluoroscopy. The participant's worst score (i.e. largest) across these three task repetitions will be recorded at each timepoint and the difference across timepoints will be calculated.
Time Frame: Post treatment (4 weeks) compared to pre-treatment baseline
Measure: Mean (Standard Deviation); unit: percentage of the C2-4 anatomical scalar
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
percentage of the C2-4 anatomical scalar | -.12 (2.5)

4. Primary Outcome: Change in Total Pharyngeal Residue Thin Liquids
Description: A videofluoroscopic measure of the amount of residue left behind in the pharynx after a swallow. This measure is obtained from pixel-based measures of the area of residue in the pharynx on a lateral view x-ray image at the end of the swallow. The number of pixels is divided by an anatomical reference scalar defined by the squared length of the distance, in pixels, between the anterior inferior corners of the C2 and C4 cervical vertebrae on the same image. The investigators will measure pharyngeal residue across a series of 3 thin liquid swallows in videofluoroscopy. The participant's worst score (i.e. largest) across these three task repetitions will be recorded at each timepoint and the difference across timepoints will be calculated.
Time Frame: Post treatment (4 weeks) compared to pre-treatment baseline
Measure: Mean (Standard Deviation); unit: percentage of the C2-4 anatomical scalar
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
percentage of the C2-4 anatomical scalar | -.24 (1.29)

5. Primary Outcome: Change in Time-to-laryngeal-vestibule-closure Mildly Thick Liquids
Description: The time interval (in milliseconds) measured on a videofluoroscopic x-ray of swallowing between onset of the hyoid burst movement at the beginning of a swallow and achieving airway protection via closure of the laryngeal vestibule. The investigators will measure time-to-laryngeal-vestibule-closure across a series of 3 mildly thick liquid swallows in videofluoroscopy. The participant's worst score (i.e. longest) across these 3 task repetitions will be recorded at each timepoint and the difference across timepoints will be calculated.
Time Frame: Post treatment (4 weeks) compared to pre-treatment baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
milliseconds | 33 (198)

6. Primary Outcome: Change in Penetration-Aspiration Scale Score Mildly Thick Liquids
Description: The Penetration-Aspiration Scale is an 8-point ordinal scale, measured on a videofluorosopic x-ray of swallowing, which documents the depth of any airway invasion events, and the subsequent response to airway invasion (Rosenbek et al., 1996). The scale ranges from a minimum score of 1 (no airway invasion) to a maximum score of 8 (entry of material below the true vocal folds with no response and no ejection). Higher scores are worse. The investigators will measure penetration-aspiration across a series of 3 mildly thick liquid swallows in videofluoroscopy. The participant's worst score (i.e. highest) across these three task repetitions will be recorded at each timepoint and the difference across timepoints will be calculated.
Time Frame: Post treatment (4 weeks) compared to pre-treatment baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
score on a scale | -1 (2)

7. Primary Outcome: Change in Pharyngeal Area at Maximum Constriction Mildly Thick Liquids
Description: A videofluoroscopic measure of the degree of pharyngeal constriction during swallowing (i.e. maximum obliteration of the space in the pharynx). This measure is obtained from pixel-based measures of the unobliterated area of the pharynx on a lateral view x-ray image at the point of maximum constriction. The number of pixels is divided by an anatomical reference scalar defined by the squared length of the distance, in pixels, between the anterior inferior corners of the C2 and C4 cervical vertebrae on the same image. The investigators will measure pharyngeal area at maximum constriction across a series of 3 mildly thick liquid swallows in videofluoroscopy. The participant's worst score (i.e. largest) across these three task repetitions will be recorded at each timepoint and the difference across timepoints will be calculated.
Time Frame: Post treatment (4 weeks) compared to pre-treatment baseline
Measure: Mean (Standard Deviation); unit: percentage of the C2-4 anatomical scalar
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
percentage of the C2-4 anatomical scalar | .28 (1.5)

8. Primary Outcome: Change in Total Pharyngeal Residue Mildly Thick Liquids
Description: A videofluoroscopic measure of the amount of residue left behind in the pharynx after a swallow. This measure is obtained from pixel-based measures of the area of residue in the pharynx on a lateral view x-ray image at the end of the swallow. The number of pixels is divided by an anatomical reference scalar defined by the squared length of the distance, in pixels, between the anterior inferior corners of the C2 and C4 cervical vertebrae on the same image. The investigators will measure pharyngeal residue across a series of 3 mildly thick liquid swallows in videofluoroscopy. The participant's worst score (i.e. largest) across these three task repetitions will be recorded at each timepoint and the difference across timepoints will be calculated.
Time Frame: Post treatment (4 weeks) compared to pre-treatment baseline
Measure: Mean (Standard Deviation); unit: percentage of the C2-4 anatomical scalar
Arm/Group | Effortful Swallow Maneuver
Number analyzed (Participants) | 5
percentage of the C2-4 anatomical scalar | -.5 (1.07)

ADVERSE EVENTS:
Time Frame: During the time frame between baseline and post 4-week treatment
Arm/Group | Effortful Swallow Maneuver
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT05319795/Prot_SAP_000.pdf